CLINICAL TRIAL: NCT01632072
Title: The Undernourished Patient: Prevention and Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Godthaab rehabilitation centre (Unknown)
Responsible Party: Principal Investigator, Per Ole Iversen, MD, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012/928
Record Dates: First submitted 2012-06-28; First posted 2012-06-29 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — Nutritional Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional counseling (Experimental): Dietary supplement
  Interventions: Dietary Supplement: Nutritional support
- No nutritional counceling (No Intervention)

INTERVENTIONS:
Dietary Supplement: Nutritional support — Nutritional support and counseling
  Arms: Nutritional counseling

SUMMARY:
The purpose of this study is to determine whether a nutrition intervention during a rehabilitation stay followed by nutritional advice after discharge, can improve the nutritional status of the patients after 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. In risk of undernutrition or undernourished according to the screening tool NRS-2002, score 3 or above.
2. Living in Oslo, Bærum or Asker municipality.
3. Must be able to cooperate.

Exclusion Criteria:

1. Unwilling to participate
2. Less than 12 months life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Body weight change | Baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Per O Iversen, MD, Principal Investigator — University of Oslo
Locations (1):
- Godthaab rehabilitation center, Bekkestua, Norway

REFERENCES:
- [Derived] Andersson J, Hulander E, Rothenberg E, Iversen PO. Effect on Body Weight, Quality of Life and Appetite Following Individualized, Nutritional Counselling to Home-Living Elderly after Rehabilitation - An Open Randomized Trial. J Nutr Health Aging. 2017;21(7):811-818. doi: 10.1007/s12603-016-0825-8. PMID 28717811
- See also: Published paper — https://www.ncbi.nlm.nih.gov/pubmed/?term=Ole+Iversen+P